CLINICAL TRIAL: NCT05828082
Title: A Phase 2 Study of M1774 in Refractory SPOP-Mutant Prostate Cancer
Brief Title: Testing the Effect of M1774 on Hard-to-Treat Refractory SPOP-mutant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-03150; NCI-2023-03150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10603 (Other: Dana-Farber - Harvard Cancer Center LAO); 10603 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2023-04-22; First posted 2023-04-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Castration-Resistant Prostate Carcinoma; Refractory Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tuvusertib) (Experimental): Patients receive tuvusertib PO QD on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, MRI, CT, PET/MRI, PET/CT or U/S and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Tuvusertib; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/MRI or PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Tuvusertib — Given PO
  Other Names: ATR Kinase Inhibitor M1774; M 1774; M-1774; M1774
Procedure: Ultrasound Imaging — Undergo U/S
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase II trial tests how well M1774 works in treating patients with prostate cancer that does not respond to treatment (refractory) and that has a mutation in the gene responsible for making the speckle type BTB/POZ protein (SPOP). M1774 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving M1774 may be able to shrink or stabilize refractory SPOP-mutant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the response rate of the ATR inhibitor tuvusertib (M1774) in highly refractory prostate cancer.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival (OS) of refractory SPOP-mutant prostate cancer patients receiving M1774.

II. To evaluate the progression-free survival (PFS) of refractory SPOP-mutant prostate cancer patients receiving M1774.

III. To evaluate the Common Terminology Criteria for Adverse Events (CTCAE) 5.0-defined adverse event (AE) rates of refractory SPOP-mutant prostate cancer patients receiving M1774.

EXPLORATORY OBJECTIVE:

I. To determine changes in SPOP-mutant circulating tumor deoxyribonucleic acid (ctDNA); SPOP-mutant prostate cancer-derived exosomes, and SPOP-, ATR-, and ATM-related gene signature changes on ATR inhibition, including RAC1, FDFT1, DHCR24, DHCR7, and MVD.

OUTLINE:

Patients receive tuvusertib orally (PO) every day (QD) on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, magnetic resonance imaging (MRI), computed tomography (CT), positron emission tomography (PET)/MRI, PET/CT or ultrasound (U/S) and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Presence of SPOP mutations in prostate cancer cells, as indicated by Next Generation Sequencing (NGS)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* Castrate-range testosterone (=< 50 ng/dL) after androgen deprivation therapy (ADT) or orchiectomy
* Prior treatment with second generation anti-androgen (2GAA) and taxane- or lutetium-based therapy. More than one kind of prior treatment with 2GAA and taxane - or lutetium-based therapies is also acceptable
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M1774 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) =< 3 x institutional upper limit of normal (ULN)
* Creatinine =< 1.5 × ULN
* Creatinine clearance >= 60 mL/min

  * Creatinine clearance should be measured if estimated glomerular filtration rate (eGFR) is > 60 mL/min
* Hemoglobin >= 9.0g/dL
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of M1774 on the developing human fetus are unknown. For this reason and because ATR inhibitors may be teratogenic (Musson et al., 2022), women of child-bearing potential who are partners of men enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to the study, for the duration of study participation, and 6 months after completion of M1774 administration. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Men enrolled on this study must agree to use adequate contraception prior to study entry, for the duration of study participation, and 3 months after completion of M1774 administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with uncontrolled intercurrent illness
* Patients who cannot discontinue proton pump inhibitors (PPIs). H2 receptor antagonists will not be permitted within 12 hours before dosing of M1774 and until 2 hours after dosing of M1774. Antacids will not be permitted within 2 hours before and 2 hours after administration of M1774
* Patients who cannot discontinue drugs that are strong inhibitors of CYP3A4 or CYP1A2
* Patients who cannot discontinue drugs that are hMATE1 or hMATE2-Ksubstrates
* Patients with a baseline QC interval > 470 msec

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Response rate | Assessed up to 6 months from trial registration
  Defined by the Prostate Cancer Working Group 3.0 criteria. Simon's two-stage design will be used.

SECONDARY OUTCOMES:
Overall Survival | From trial registration until death due to any cause, assessed up to 2 years
  From trial registration until death due to any cause
Progression Free Survival (PFS) | From trial registration until the first indication of disease progression (or death), assessed up to 2 years
  The median PFS time, as well as a 95% confidence interval, will be constructed using the Kaplan-Meier method.
Incidence of adverse events (AE) | Up to 2 years from registration date
  Maximum grade AE's will be summarized using simple counting statistics in a tabular fashion. This will be done both with and without regard to treatment attribution. Will be assessed using Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Overall SPOP-driven gene signature changes | At cycle 1, day 9 and time of progression
  Overall SPOP-driven gene signature changes over the course of treatment will be measured by ribonucleic acid sequencing. These will include SPOP targets RAC1, FDFT1, DHCR24, DHCR7, and MVD. Changes in expression over time will be compared using a Wilcoxon signed-rank test. Changes in circulating SPOP-mutant fraction of circulating tumor deoxyribonucleic acid in responders will be compared to changes in non-responders using Student's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Orme, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (26):
- United States (26):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT05828082/ICF_000.pdf